CLINICAL TRIAL: NCT02077647
Title: A Focused Registry on the Conservative Treatment of Osteoarthritis of the Knee
Brief Title: Focused Registry on the Conservative Treatment of Osteoarthritis of the Knee
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FR_Tomofix
Record Dates: First submitted 2014-02-12; First posted 2014-03-04 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis, Knee; Osteonecrosis
Keywords: Knee osteoarthritis; knee osteonecrosis; osteotomy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Conservative: Conservative treatment of osteoarthritis of the knee

SUMMARY:
The primary objective of this registry is to assess the functional outcome measured with the Knee Injury and Osteoarthritis Outcome Score (KOOS) for patients with medial unicompartmental osteoarthritis and osteonecrosis of the knee treated conservatively. The aim of the Focused Registry is to complete the data collection and enable a sound analysis for the Tomofix Small size study.

DETAILED DESCRIPTION:
The aim of the Focused Registry is to complete the data collection and enable a sound analysis for the Tomofix Small size study.

The incidence of knee osteoarthritis (OA) is higher in Japan than in other populations. Respective prevalences of 47.0 and 70.2% in men and women for Kellgren-Lawrence Grades 2-4 knee OA are reported in Japanese patients aged 60 years and over.

First treatment options are pharmacological (i.e. NSAIDs) and non-pharmacological therapies (i.e. use of assistive devices, exercises, osteopathy, physical therapy), followed by injections of hyaluronic acid and other substances. If no such therapies are successful, surgical treatment options as unicompartmental knee replacement, total knee arthroplasty and high tibial osteotomy (HTO) are recognized. The discussion of which is the best therapy is still controversial. HTO may decrease the number of complications compared to total knee replacement or unicompartmental knee arthroplasty and leave the option for later replacement surgery.

In this project, patients are included who would be surgically treated with HTO with Tomofix small based on the investigator's assessment but refuse to have surgical treatment. They will be treated conservatively and are investigated to serve as reference to an ongoing clinical study investigating invasive treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older
* Patients with OA Grade 1-4 (Kellgren-Lawrence) or osteonecrosis (ON) Stage 2-4 (according to the Koshino classification)
* Indication for open wedge HTO with the TomoFix™ Small
* No ligamental laxity
* Able to understand and read country national language at an elementary level
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the registry according to the registry plan (RP)
* Signed and dated IRB/EC-approved written informed consent

Exclusion Criteria:

* Femoro-tibial angle (FTA) > 190° (standing view x-ray)
* Flexion contracture > 15°
* Total knee replacement or unicompartmental knee on the contralateral side
* Infections located between the middle of the femur and the ankle
* Systemic bacterial infections
* Severe osteoarthritis or surgery of the hip joint
* Smoking of more than 20 cigarettes per day
* Immunodeficiency or compromised host
* Patients who have participated in any other device or drug related clinical trial within the previous month
* ACL/PCL reconstruction of the same knee
* Severe osteoarthritis of the ipsilateral ankle joint
* HTO on the contralateral side
* Major surgery on both knees (minor surgery as arthroscopic meniscectomy and synovectomy is allowed)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Indication for open wedge HTO with the TomoFix™ Small presenting in the orthopaedic department of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Function of the knee | 24 months
  Knee Injury and Osteoarthritis Outcome Score (KOOS)

SECONDARY OUTCOMES:
Patient-evaluated function of the knee and quality of life | 6 months, 12 months, 24 months
  Oxford-12-item knee score, WOMAC (as calculated from the KOOS)
Clinician-evaluated function of the knee | 6 months, 12 months, 24 months
  Japanese Orthopaedic Association (JOA) score
Health-related quality of life | 6 months, 12 months, 24 months
  Short Form-36 (SF-36)
Range of motion (ROM) | 6 months, 12 months, 24 months
Local and general pain | 6 months, 12 months, 24 months
  Visual Analogue Scale (VAS)
Possibility and duration of the Japanese sitting style | 6 months, 12 months, 24 months
Return to sport activities | 6 months, 12 months, 24 months
Utilization | up to hospital discharge
  Length of hospital stay
Evaluation of degenerated and regenerated cartilage | intraoperative and after 2 years
  ICRS and Outerbridge / Koshino)
Radiological parameters | 6 months, 12 months, 24 months
  Kellgren-Lawrence classification, joint space narrowing, tibial slope, tibia vara
Complications | 6 months, 12 months, 24 months
  Complications due to injections, complications due to heat therapy, complications due to medication (NSAIDs)
Anatomical alignment | 6 months, 12 months, 24 months
  Femoro tibial angle (FTA)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Faeh, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland; Takeshi Sawaguchi, MD, Principal Investigator — Toyama Municipal Hospital, Toyama-city, Japan
Locations (4):
- Japan (4):
  - Nagasaki University, Nagasaki
  - Osaka Koseinenkin Hospital, Osaka
  - Hashiba Orthopaedic Clinic, Toyama
  - Toyama Municipal Hospital, Toyama

REFERENCES:
- [Background] Takeuchi R, Aratake M, Bito H, Saito I, Kumagai K, Hayashi R, Sasaki Y, Akamatsu Y, Ishikawa H, Amakado E, Aota Y, Saito T. Clinical results and radiographical evaluation of opening wedge high tibial osteotomy for spontaneous osteonecrosis of the knee. Knee Surg Sports Traumatol Arthrosc. 2009 Apr;17(4):361-8. doi: 10.1007/s00167-008-0698-4. Epub 2009 Jan 23. PMID 19165468
- [Background] Takeuchi R, Ishikawa H, Aratake M, Bito H, Saito I, Kumagai K, Akamatsu Y, Saito T. Medial opening wedge high tibial osteotomy with early full weight bearing. Arthroscopy. 2009 Jan;25(1):46-53. doi: 10.1016/j.arthro.2008.08.015. Epub 2008 Oct 10. PMID 19111218
- [Background] Takeuchi R, Saito T, Koshino T. Clinical results of a valgus high tibial osteotomy for the treatment of osteoarthritis of the knee and the ipsilateral ankle. Knee. 2008 Jun;15(3):196-200. doi: 10.1016/j.knee.2008.02.002. Epub 2008 Mar 25. PMID 18367399